CLINICAL TRIAL: NCT03080077
Title: Safety and Effectiveness of Corneal Crosslinking (CXL): Keratoconus and Post-Refractive Ectasia
Acronym: CXL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Penny Asbell, Professor of Ophthalmology, Director of Cornea and Refractive Services, Director of the Cornea Fellowship Program, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 16-0627
Record Dates: First submitted 2017-03-06; First posted 2017-03-15 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Keratoconus; Ectasia
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic | interventions — Iontophoresis; Corneal Cross-Linking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epi-Off CXL (Active Comparator): Using topical anesthesia (proparacaine), the surgeon will create a complete corneal abrasion to facilitate riboflavin diffusion into the cornea. The epithelium will be removed by gently brushing the cornea with a scalpel. A corneal abrasion diameter of ~9mm is recommended, which may be adjusted as needed at the discretion of the investigator to accommodate individual eye geometry. Ultrasound corneal pachymetry should be performed before dis-epithelialization and after dis- epithelialization. Local anesthetics will be administered as needed to maintain patient comfort during the CXL procedure.
  Interventions: Drug: Epi-Off
- Epi-On CXL (Experimental): The IONTOPHOR CXL iontophoresis applicator and the associated blepharostat will be placed onto the cornea to be treated. The applicator will be secured to the cornea and filled with Ricrolin+ which as been aspirated from the bottle using a syringe with a needle. The generator will be switched on and set to 1 mA for 5 minutes. The generator will then be disconnected and the applicator will be removed from the cornea.
  Interventions: Drug: Ricrolin+

INTERVENTIONS:
Drug: Ricrolin+ — The IONTOPHOR CXL iontophoresis applicator and the associated blepharostat will be placed onto the cornea to be treated. The applicator will be secured to the cornea and filled with Ricrolin+ which as been aspirated from the bottle using a syringe with a needle. The generator will be switched on and set to 1 mA for 5 minutes. The generator will then be disconnected and the applicator will be removed from the cornea.
  Other Names: Epi-on (iontophoresis)
  Arms: Epi-On CXL
Drug: Epi-Off — Using topical anesthesia (proparacaine), the surgeon will create a complete corneal abrasion to facilitate riboflavin diffusion into the cornea. The epithelium will be removed by gently brushing the cornea with a scalpel. A corneal abrasion diameter of ~9mm is recommended, which may be adjusted as needed at the discretion of the investigator to accommodate individual eye geometry. Ultrasound corneal pachymetry should be performed before dis-epithelialization and after dis- epithelialization. Local anesthetics will be administered as needed to maintain patient comfort during the CXL procedure.
  Arms: Epi-Off CXL

SUMMARY:
This prospective, randomized study is being conducted to evaluate the safety and effectiveness of corneal cross-linking (CXL) in patients with keratoconus or post-refractive ectasia (post-LASIK or PRK) utilizing two techniques: the "standard" Epi-Off technique or an Epi-On technique that utilizes iontophoresis (I-CXL) to deliver the riboflavin to the cornea without need for removal of the corneal epithelium. Patients will be randomized to receive CXL treatment with either the Epi-On or Epi-Off technique.

ELIGIBILITY:
Inclusion:

1. 10 years of age or older
2. Understand and have signed written IRB-approved informed consent
3. Willingness and ability to comply with schedule for follow-up visits
4. Having a diagnosis of keratoconus or post-refractive corneal ectasia (post-LASIK or PRK)
5. Presence of central or inferior steepening on the Pentacam map
6. Axial topography consistent with keratoconus or post-refractive corneal ectasia (post-LASIK or PRK)
7. Presence of one or more slit lamp findings associated with keratoconus, such as:

   1. Scissoring of the retinoscopic reflex
   2. Fleischer ring
   3. Vogt striae
   4. Corneal thinning
   5. Corneal scarring
8. BSCVA 20/20 or worse (<58 letters on ETDRS chart).
9. Contact lens wearers only: Removal of contact lenses for the required period of time prior to the first refraction:

Contact Lens Type Minimum Discontinuation Time Soft 3 Days Soft Extended Wear 1 Week Soft Toric 2 Weeks Rigid gas permeable 2 Weeks Hybrid lenses (SynergEyes; Rose K; Clear Kone) 2 Weeks Scleral Lenses 2 Weeks

Exclusion Criteria: All subjects meeting any of the following criteria will be excluded from the study:

1. A history of previous corneal surgery in the eye to be treated (including previous CXL treatment)

   a. Eyes with episodes of hydrops or scarring from hydrops may be included as long as there is no active inflammation
2. Corneal pachymetry < 400 microns at the thinnest point measured by Pentacam
3. Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications or prevent the possibility of improved vision, for example:

   1. History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, corneal melt, or corneal dystrophy, etc.)
   2. Clinically significant corneal scarring in the treatment zone
4. A history of chemical injury or delayed epithelial healing in the eye(s) to be treated
5. Pregnancy (including plan to become pregnant) or lactation during the procedure
6. A known sensitivity to study medications
7. Nystagmus or any other condition that would prevent a steady gaze during the cross-linking treatment or other diagnostic tests
8. A condition that, in the investigator's opinion, would interfere with or prolong epithelial healing
9. Presence or history of any other condition or finding that, in the investigator's opinion, makes the patient unsuitable as a candidate for cross-linking or study participation or may confound the outcome of the study
10. Inability to cooperate with diagnostic tests or inability to understand the informed consent.
11. Concurrent use of systemic (including inhaled) medications that may impair healing, including but not limited to: antimetabolites, isotretinoin (Accutane®) within 6 months of treatment, and amiodarone hydrochloride (Cordarone®) within 12 months of treatment.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change in Kmax | baseline and 2 years
  Kmax = maximum simulated keratometry value

SECONDARY OUTCOMES:
Change in steepest K | baseline and 2 years
  steepest K is the higher diopter number which represents the steepest meridian of the cornea
Change in astigmatism | baseline and 2 years
  Astigmatism is an imperfection in the curvature of the cornea, causing a refractive error diagnosed by standard eye exam with refraction test.
Change in keratometry | baseline and 2 years
  Keratometry is the measurement of the corneal radius of curvature
Change in pachymetry | baseline and 2 years
  Pachymetry is a common test for glaucoma and measures the thickness of the cornea
Changes in curvature | baseline and 2 years
  Shape of cornea
Change in sphere | baseline and 2 years
  Change in refraction
Change in cylinder | 2 years
  Cylinder is the amount of astigmatism that is present
Change in BCVA | baseline and 2 years
  Best-corrected visual acuity (BCVA)

CONTACTS AND LOCATIONS:
Overall Officials: Penny A Asbell, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lombardo M, Serrao S, Rosati M, Ducoli P, Lombardo G. Biomechanical changes in the human cornea after transepithelial corneal crosslinking using iontophoresis. J Cataract Refract Surg. 2014 Oct;40(10):1706-15. doi: 10.1016/j.jcrs.2014.04.024. PMID 25263041
- [Background] Koller T, Schumacher S, Fankhauser F 2nd, Seiler T. Riboflavin/ultraviolet a crosslinking of the paracentral cornea. Cornea. 2013 Feb;32(2):165-8. doi: 10.1097/ICO.0b013e318269059b. PMID 23187160